CLINICAL TRIAL: NCT05316298
Title: Gentamicin-loaded Calcium Sulfate-hydroxyaPatite Biocomposite to tREat Diabetic Foot Ulcers Complicated by oSteomyElitis: a pRospectiVE Cohort Study
Brief Title: Diabetic Foot Osteomyelitis Treatment Using Gentamicin-loaded Calcium Sulfate-hydroxyapatite Biocomposite
Acronym: PRESERVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Ziekenhuisgroep Twente (Other); Slingeland Hospital (Other); Franciscus Gasthuis (Other); UMC Utrecht (Other); Rijnstate Hospital (Other); Jeroen Bosch Ziekenhuis (Other); Reinier de Graaf Groep (Other); St. Antonius Hospital (Other); St Jansdal Hospital (Other); Maasstad Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200240
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Foot Ulcer; Osteomyelitis; Diabetes Mellitus
Keywords: Surgical treatment; antibiotic-loaded bone graft substitute; Cerament G
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PRESERVE protocol: Treatment according to the PRESERVE protocol consists of 2 study phases. Phase 1 consists of standard-of-care non-surgical treatment, performed in accordance with current treatment guidelines, during which the research team performs observations.
  After failed standard-of care non surgical treatment, subjects will be included in study phase 2 and undergo treatment by surgical debridement of the diabetic foot ulcer and underlying osteomyelitis, followed by bone void filling with gentamicin-loaded calcium sulfate-hydroxyapatite biocomposite and closure of soft tissues and skin, followed by postoperative treatment regimen including woundcare, 10 days of antibiotics and offloading.

SUMMARY:
The amputation risk is high when diabetic foot ulcers, complicated by osteomyelitis, fail to heal after non-surgical standard-of-care treatment. A new treatment regimen has been developed recently and has been proven feasible. This treatment regimen consists of surgical debridement, followed by bone void filling with gentamicin-loaded calcium sulfate-hydroxyapatite biocomposite and closure of soft tissues and skin, in combination with antibiotic therapy and offloading. This treatment regimen has not been investigated prospectively.

Therefore, this multicenter prospective cohort study was designed, with the primary objective of investigating postoperative wound healing. Patients with diabetic forefoot ulcers, complicated by osteomyelitis, will be included. The most relevant exclusion criteria are: Severe diabetic foot infection, severe limb ischemia, and foot deformity causing high pressure and friction on the diabetic foot ulcer. After inclusion, subjects will undergo study phase 1, which is observation of the standard-of-care non-surgical treatment. When standard-of-care non-surgical treatment is unsuccessful, subjects will be included in study phase 2, which consists of treatment by surgical debridement of the diabetic foot ulcer and underlying osteomyelitis, followed by bone void filling with gentamicin-loaded calcium sulfate-hydroxyapatite biocomposite and closure of soft tissues and skin, followed by a postoperatieve treatment regimen which involves wound care, 10 days of antibiotic therapy and offloading.

The primary outcome measure of this study is the proportion of subjects with post-operative wound healing, which will be investigated clinically and will be objectified by a review panel of blinded, independent experts based on digital photographs. Follow-up will be performed until wound healing or for a maximum of 20 weeks. The primary outcome measure is the proportion of subjects with postoperative wound healing during 20 weeks of follow-up. Secondary outcome measures are: days until postoperative wound healing, proportion of subjects with persistent osteomyelitis post-operatively, proportion of subjects undergoing amputations during follow-up, foot function index scores at inclusion and after 20 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* One or multiple forefoot diabetic foot ulcers complicated by osteomyelitis. The treating physician will diagnose osteomyelitis, based on either positive culture results or histopathologic findings of a bone sample, or on the combination of clinical findings of inflammation and a positive probe-to-bone test or imaging findings (X-ray, MRI) A patient with multiple forefoot DFOs can be included as long as all ulcers are related to osteomyelitis on one location.
* Sufficient soft tissues and skin for primary closure or closure by local tissue transposition after surgical debridement, as judged by the treating physician.
* Written declaration of informed consent

Exclusion Criteria:

* Acute Charcot neuroarthropathy, which will be diagnosed by the treating physician based on clinical examination and MRI.
* Adequate surgical debridement is possible by performing an amputation, as judged clinically by the treating physician (e.g. DFO on the 4th or 5th digit).
* Contra-indications for the use of gentamicin-loaded calcium sulfate-hydroxyapatite biocomposite, as mentioned by the producer: hypersensitivity to any aminoglycoside antibiotics, myasthenia gravis, severe renal impairment, pre-existing calcium metabolism disorders, pregnancy, and breastfeeding. This information will be investigated using the patient's electronic health record file and verbal verification. Severe renal impairment is defined as chronic kidney disease with an estimated glomerular filtration rate <30 ml/min/1.73m2 or renal replacement therapy.
* Foot deformities that lead to increased pressure and friction on the site of the ulcer, which can only be adequately managed by surgical correction, as judged clinically by the treating physician.
* Implants in bone affected by osteomyelitis
* Inadequate quality and / or volume of soft tissues and skin for primary closure or closure by local tissue transposition after surgical debridement, as judged by the treating physician.
* No written declaration of informed consent.
* Osteomyelitis on ≥1 separate locations.
* Other infected diabetic foot ulcers.
* Severe chronic limb Ischemia, defined in accordance with the Wound-, Ischemia-, Foot Infection classification as signs and / or symptoms of peripheral artery disease and a systolic toe pressure < 30 mmHg and/or a transcutaneous oxygen pressure < 30 mmHg in the forefoot.Previous revascularisation is no exclusion criterion.
* Severe communication disabilities as judged by the treating physician, which would interfere with adherence to instructions.
* Severe diabetic foot infection, defined as infection-grade 4 according to the International Working Group on the Diabetic Foot classification.
* Severely immunocompromised state as judged by the treating physician (e.g., neutropenia due to chemotherapy, high doses of corticosteroids, HIV infection with CD4 count <200 / µl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, patients will be included who present in one of the 10 participating Dutch hospitals with forefoot diabetic foot ulcers complicated by osteomyelitis and sufficient skin and soft tissues around the ulcer for surgical closure.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative wound healing | 20 weeks
  Macroscopic complete epithelialization of all surgical wounds after removal of sutures and/or staples without drainage for a minimum of 2 weeks.

SECONDARY OUTCOMES:
Duration to postoperative wound healing | 20 weeks
  Duration to postoperative wound healing, expressed in days postoperatively.
persistent osteomyelitis postoperatively | 20 weeks
  The proportion of subjects without postoperative wound healing and with persistent osteomyelitis, diagnosis based on clinical findings (signs of inflammation) in combination with suggestive findings of osteomyelitis on imaging (X-ray, MRI) or a positive probe-to-bone test.
Amputations during follow-up | 20 weeks
  Proportion of patients undergoing amputations (minor = distal to the ankle joint, major = proximal to the ankle joint)
Foot Function Index (FFI) scores | 20 weeks
  Pre-operatively and at final follow-up, subjects will fill-in FFI-5pt questionnaires. These consist of 15 questions regarding pain in the foot and functional problems due to foot problems. These are translated in Dutch and have previously been validated. We will calculate the overall FFI scores and those or the domains of 'pain' and 'disability'. Per patient, we will also calculate the changes in mean or median FFI-5pt scores overall and separately for the domains of 'pain' and 'disability', by subtracting the FFI-5pt score measured at final follow-up from the FFI-5pt score measured at inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Kor H. Hutting, M.D., Principal Investigator — University Medical Center Groningen
Locations (10):
- Netherlands (10):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Hospitalgroup Twente, Almelo
  - Rijnstate Hospital, Arnhem
  - Reinier de Graaf Hospital, Delft
  - Slingeland Hospital, Doetinchem
  - St. Jansdal Hospital, Harderwijk
  - St. Antonius Hospital, Nieuwegein
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Maasstad Hospital, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study the data will be made publically available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Expected to become available in june 2024 for 10 years.
Access Criteria: Upon requrest by a professional researcher with a valid research plan.